CLINICAL TRIAL: NCT00601978
Title: A 12-Week, Multi-center, Randomized, Prospective, Open-Label, Blinded Rater, Crossover Study of the Effects of Immediate-Release Carbidopa/Levodopa Versus Carbidopa/Levodopa/Entacapone on Markers of Event-Related Potentials (ERPs) in Patients With Idiopathic Parkinson's Disease and End-of-Dose Wearing Off
Brief Title: Carbidopa/Levodopa Versus Carbidopa/Levodopa/Entacapone on Markers of Event Related Potentials (ERPs) in Patients With Idiopathic Parkinson's Disease (PD) and End-of-dose Wearing Off
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision brand strategy; no patients enrolled
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CELC200AUS15
Record Dates: First submitted 2008-01-11; First posted 2008-01-28 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; carbidopa/levodopa/entacapone; carbidopa/levodopa; non-motor symptoms; event-related potential; ERP; EEG; electroencephalogram
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Stalevo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Immediate-Release Carbidopa/Levodopa
  Interventions: Drug: carbidopa/levodopa
- 2 (Active Comparator): Carbidopa/Levodopa/Entacapone
  Interventions: Drug: Carbidopa/Levodopa/Entacapone

INTERVENTIONS:
Drug: carbidopa/levodopa
  Arms: 1
Drug: Carbidopa/Levodopa/Entacapone
  Other Names: Stalevo
  Arms: 2

SUMMARY:
This study will evaluate the effects of immediate release (IR) carbidopa levodopa versus the effects of immediate-release carbidopa/levodopa on ERP parameters in patients with idiopathic PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 45 to 75 years (inclusive)
2. Patients with an MMSE score of at least 25 at the screening visit.
3. Patients who experience EODWO, which is the re-emergence of PD symptoms during the waking hours, as determined by a WOQ-9 score of at least one motor symptom of wearing off
4. Patients taking a stable dose of immediate-release carbidopa/levodopa for at least 4 weeks prior to randomization, at an equivalent total daily dose of levodopa between 300 to 600 mg/day.
5. Patients who, in the investigator's judgement, are capable of satisfying the requirements of the protocol
6. Patients who are willing and able to give written informed consent according to legal requirements.

Exclusion Criteria:

1. Diagnosis of secondary parkinsonism, atypical Parkinson's disease, or history, signs, or symptoms suggesting these diagnoses.
2. Unstable Parkinson's disease as determined by the investigator.
3. Disabling dyskinesia (a score of >2 on the Unified Parkinson's Disease Rating Scale [UPDRS] question #32, or a score of >2 on UPDRS question #33).
4. Treatment with carbidopa/levodopa controlled-release or extended-release formulations (bedtime administration is acceptable). The use of controlled-release carbidopa/levodopa is not allowed on the evening before the visits in which efficacy assessments occur.
5. Concomitant or previous treatment with certain medications or supplements as specified in the protocol.
6. Patients who are unable to comply with the dosing requirements of the protocol, such that the first dose of study medication will be taken after the time of the first EEG and the second dose will be taken after completion of the third EEG.
7. Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR; diagnosis of 1. dementia (of any cause); 2. moderate or severe major depression, present independent from the time of first diagnosis of PD, as defined by a QIDS-SR16 score of > 15; or 3. generalized anxiety disorder or panic disorder if made prior to the diagnosis of PD.
8. DSM-IV-TR diagnosis of alcohol or substance abuse (excluding nicotine or caffeine) during the 3 months prior to randomization) or alcohol or substance dependence (excluding nicotine or caffeine) during the 6 months prior to randomization. Alcohol should be avoided within the 12 hours preceding the Week 6 and Week 12 visits.
9. Nicotine use of >5 cigarettes (or equivalent in other forms of administration) per day. Nicotine use will not be permitted on the day of the Week 6 and Week 12 visits.
10. Ingestion of >4 caffeinated beverages (or equivalent in other forms of administration) per day.
11. History of major head injury, including skull fracture or a penetrating head injury, or a history of brain surgery.
12. Past or current treatment by deep brain stimulation.
13. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
14. Hearing loss or impairment that may prevent reliability of test results using auditory evoked potentials.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the mean latency of the P300 component of the event-related potentials (ERPs) at four hours post study-drug administration

SECONDARY OUTCOMES:
Mean latency of the P300 component of ERPs at pre-dose and 1 hours post-dose study drug administration
Mean latency of the N100 component of ERPs at pre-dose, 1 hour post-dose and 4 hours post-dose study drug administration
Pharmacokinetics at 9.25 and 12.55 hours post dose